CLINICAL TRIAL: NCT01518166
Title: A Two-way Cross-over, Placebo-controlled Interaction Trial in Two Parts (in Healthy Subjects), Studying Liraglutide's Potential Influence on the Absorption Pharmacokinetics of Lisinopril, Atorvastatin, Griseofulvin and Digoxin, and Liraglutide's Potential Influence on Intragastric pH
Brief Title: Effect of Liraglutide on Gastrointestinal Absorption of Several Drugs and Potential Influence of Liraglutide on Intragastric pH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1608; 2006-000175-15 (EudraCT Number)
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide; Atorvastatin; Lisinopril; Griseofulvin; Digoxin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial period A (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo; Drug: atorvastatin; Drug: lisinopril
- Trial period B (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo; Drug: griseofulvin; Drug: digoxin

INTERVENTIONS:
Drug: liraglutide — Administered as a subcutaneous injection. Initial dose 0.6 mg daily, adjusted to 1.2 mg daily in week 2 and escalated to 1.8 mg daily in week 3
Drug: placebo — Administered as a subcutaneous injection. Given as daily volume of 100 mcl, 200 mcl and 300 mcl respectively
Drug: atorvastatin — One single dose of 40 mg. Tablet
  Arms: Trial period A
Drug: lisinopril — One single dose of 20 mg. Tablet
  Arms: Trial period A
Drug: griseofulvin — One single dose of 500 mg. Tablet
  Arms: Trial period B
Drug: digoxin — One single dose of 1 mg. Tablet
  Arms: Trial period B

SUMMARY:
The trial is conducted in Europe. The aim of the trial is to investigate if there is any drug to drug interaction between liraglutide and atorvastatin (Lipitor®), lisinopril (Zestril®), griseofulvin and digoxin (Lanoxin®).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects if using adequate anti-contraception or is sterile
* Body Mass Index (BMI) of 18-30 kg/m^2 (both inclusive)
* Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs and blood and urinary laboratory assessments
* Willing and capable to self-administer a subcutaneous injection

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders that may interfere with the objectives of the trial, as judged by the investigator
* Impaired renal function
* Blood pressure and heart rate in supine position outside the ranges 90-140 mmHg systolic, 50-90 mmHg diastolic and heart rate 40-100 beats/min
* Any clinically significant abnormal ECG
* Active hepatitis B and/or active hepatitis C
* Positive HIV (human immunodeficiency virus) antibodies
* Known or suspected allergy to trial product(s) or related products
* Use of any prescription or non-prescription medication except for paracetamol, nasal spray or drops for nasal congestion, and vitamins within 2 weeks prior to first dosing and during the entire trial period
* History of alcoholism or drug abuse during the last 12 months
* Smoking of more than 10 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve of atorvastatin
Area under the curve of lisinopril
Area under the curve of griseofulvin
Area under the curve of digoxin

SECONDARY OUTCOMES:
Area under the curve of liraglutide
Cmax, maximum concentration
tmax, time to reach Cmax
Terminal elimination rate constant
Intragastric pH
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Uppsala, Sweden

REFERENCES:
- [Result] Malm-Erjefalt M, Ekblom M, Vouis J, Zdravkovic M, Lennernas H. Effect on the Gastrointestinal Absorption of Drugs from Different Classes in the Biopharmaceutics Classification System, When Treating with Liraglutide. Mol Pharm. 2015 Nov 2;12(11):4166-73. doi: 10.1021/acs.molpharmaceut.5b00278. Epub 2015 Oct 12. PMID 26426736
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com